CLINICAL TRIAL: NCT06846112
Title: Randomized Clinical Trial Aimed at Comparing Unclamped Robotic Partial Nephrectomy With or Without Renorrhaphy. Randomized Control Trial Comparing Off-clamp Robotic Partial Nephrectomy With or Without Renorrhaphy. Project: GR-2021-12373396
Brief Title: Randomized Clinical Trial Aimed at Comparing Unclamped Robotic Partial Nephrectomy With or Without Renorrhaphy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: RS1835/23
Record Dates: First submitted 2024-03-06; First posted 2025-02-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized trial on surgical techniques used in clinical practice, relating to patients with organ-confined renal tumors who are candidates for OCRPN surgery, designed with the aim of prospectively demonstrating that SL-ocRPN is not inferior to RR-ocRPN in terms of surgical results (expressed by the Trifecta rate)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RR-ocRPN (Experimental): Subjects assigned to group A will receive surgical treatment through robotic partial nephrectomy (RPN), through an off-clamp and sutureless approach (SL)
  Interventions: Procedure: Robotic partial nephrectomy
- SL-ocRPN (Active Comparator): Subjects assigned to group B will receive surgical treatment of robotic partial nephrectomy (RPN), through temporary closure of the renal hilar vessels and renorrhaphy (RR), i.e. by juxtaposing the resection margins of the enucleation bed
  Interventions: Procedure: Robotic partial nephrectomy

INTERVENTIONS:
Procedure: Robotic partial nephrectomy — Robotic partial nephrectomy (RPN) is the treatment of choice for organ-confined renal tumors. For to improve functional outcomes, we designed an off-clamp and suture-free approach (SL) to limit the ischemic damage and destruction of the renal parenchyma caused, respectively, by temporary closure of the vessels of the renal hilum and by renorrhaphy (RR) (i.e. by the juxtaposition of the margins of resection of the enucleation bed, which is commonly performed at the end of tumor exeresis using suture threads stopped by surgical clips)

SUMMARY:
Intended to minimize ischemia during robotic partial nephrectomy (RPN) procedures "by any means possible".

Before starting enucleation, the boundaries of the tumor are marked during SL-ocRPN surgery cautery. Once the tumor is removed, the resection bed is cauterized by dispensing monopolar energy with "quasi-contact" mode, and hemostasis is progressively improved.

DETAILED DESCRIPTION:
Since RR impacts postoperative renal function, we believe the use of cautery instead of suture of the parenchymal breach after tumor enucleation provides at least postoperative functional results not lower, shorten the intervention time and reduce the direct costs associated with the procedure.

Based on available pilot studies, SL-ocRPN is safe, fast, and both the transfusion rate and duration of the hospital stay are not affected by the lack of renorrhaphy at the end of the enucleation. At the same time, this surgical approach does not require the use of a robotic needle holder and this can result in a reduction of direct costs related to treatment.

Furthermore, based on the preliminary data available, the rate of positive surgical margins would also not result influenced by the absence of RR and the risk of local recurrence could even be reduced by the extended one coagulation of the tumor bed after enucleation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* radiological diagnosis of organ-confined renal neoplasm (cT1-2 cN0);
* patient who is a candidate, due to personal or tumor characteristics, for ocRPN intervention;
* compliant patient, able to follow the procedures/follow-up;
* patient who agrees to participate in the clinical study and the planned randomization, by signing the informed consent.

Exclusion Criteria:

* preoperative evidence of unilateral/bilateral synchronous renal neoplasms;
* personal history of renal surgery for benign or malignant pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2028-07-07 (Estimated); Study Completion 2028-07-07 (Estimated)

PRIMARY OUTCOMES:
Trifecta rate | 36 months
  The Trifecta rate [defined as negative surgical margins, no major complications, no >30% glomerular filtration rate reduction] will be assessed and used to compare outcomes in the 2 arms.
  Then prospectively demonstrate that sutureless (SL) ocRPN is non-inferior to RR ocRPN in terms of surgical outcome.

OTHER OUTCOMES:
Direct costs | 36 months
  To prospectively compare direct costs associated with ocRPN with or without RR. For the purposes of the study, the out-of-pocket costs of the study, of the robotic instruments used, will be systematically recorded and used to estimate the direct costs associated with ocRPN with or without RR and the two surgical approaches will be compared accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Brassetti, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No